CLINICAL TRIAL: NCT06118216
Title: Costal Cartilage Donor-site Pain: Does Abdominal Muscle Infiltration Analgesia Work? A Randomized Controlled Clinical Trial of Microtia Patients
Brief Title: Costal Cartilage Donor-site Pain: Does Abdominal Muscle Infiltration Analgesia Work?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaohui Su (Other)
Responsible Party: Sponsor-Investigator, Xiaohui Su, clinical physician, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCDPDAMIAW
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Rectus Abdominis and External Oblique Muscle Infiltration Analgesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-PCIA (Placebo Comparator)
  Interventions: Procedure: intravenous patient-controlled anesthesia
- Group-IA+PCIA (Experimental)
  Interventions: Procedure: rectus abdominis(RAM) and external oblique muscle(EOM) infiltration analgesia; Procedure: intravenous patient-controlled anesthesia

INTERVENTIONS:
Procedure: rectus abdominis(RAM) and external oblique muscle(EOM) infiltration analgesia — After suturing the muscular fascia, an indwelling catheter was placed above the RAM and EOM and under the subcutaneous tissue and then sutured to the skin for fixation. Approximately 30 min before surgery completion, 1 mg/kg of 0.2% ropivacaine was infused through the indwelling catheter for IA. Additionally, 1 mg/kg of 0.2% ropivacaine was infused through the indwelling catheter every 12 h, starting 8 h postoperatively, injected four times.
  Arms: Group-IA+PCIA
Procedure: intravenous patient-controlled anesthesia — After completion of the operation, the anesthesiologist used the IPCA device; it was programmed with a background infusion rate of 2 mL/h, a bolus volume of 2 mL, and a lockout interval of 15 minutes. The 100 mL total volume of the PCA consisted of normal saline, 2.0 ug/kg sufentanil, and adjuvant antiemetic (tropisetron).

SUMMARY:
Donor-site pain is an adverse effect of autologous ear reconstruction. A well-planned pain management protocol is needed. The objective of this study was to introduce rectus abdominis and external oblique muscle infiltration analgesia (RAM+EOM-IA) in autologous ear reconstruction and to evaluate its efficacy and safety.

DETAILED DESCRIPTION:
Patients were included in two cohorts: intermittent RAM+EOM-IA combined with intravenous patient-controlled anesthesia (IPCA) and IPCA alone. The primary outcome was the numerical rating score (NRS) of pain recorded during 48 h postoperatively. Secondary outcomes included the Barthel index and rescue analgesic consumption. Additionally, areas of sensory block were tested using a cold stimulus.

ELIGIBILITY:
Inclusion Criteria:

* All patients were microtia and underwent the first stage of autologous ear reconstruction by the same experienced surgeon in First Affiliated Hospital of Fujian Medical University.

Exclusion Criteria:

* Patients were excluded if they over 18 years old; discontinued analgesic therapy; regularly used opioids, other analgesics, sedative medications, or corticosteroids; were unable to express pain scores due to comorbidities such as mental retardation; or had incomplete data.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
numeric rating scale | 4,8,12,16,20,24,28,32,36,40,44,48hours after surgery
  The primary outcome was the numerical rating score (NRS) of pain recorded during 48 h postoperatively
Rescue analgesics consumption | 48hours after surgery
  Rescue analgesics were administered only on demand and not routinely. During the postoperative days, physicians prescribed 15 mg/kg oral acetaminophen if the pain was unbearable.

SECONDARY OUTCOMES:
Barthel's index | 24hours after surgery
  The Barthel's index measures the ability to perform daily activities after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Niiyama Y, Yotsuyanagi T, Yamakage M. Continuous wound infiltration with 0.2% ropivacaine versus a single intercostal nerve block with 0.75% ropivacaine for postoperative pain management after reconstructive surgery for microtia. J Plast Reconstr Aesthet Surg. 2016 Oct;69(10):1445-9. doi: 10.1016/j.bjps.2016.05.009. Epub 2016 Jun 2. PMID 27350268
- [Background] Woo KJ, Kang BY, Min JJ, Park JW, Kim A, Oh KS. Postoperative pain control by preventive intercostal nerve block under direct vision followed by catheter-based infusion of local analgesics in rib cartilage harvest for auricular reconstruction in children with microtia: A randomized controlled trial. J Plast Reconstr Aesthet Surg. 2016 Sep;69(9):1203-10. doi: 10.1016/j.bjps.2016.06.026. Epub 2016 Jul 9. PMID 27430605
- [Background] Shaffer AD, Jabbour N, Visoiu M, Yang CI, Yellon RF. Paravertebral Nerve Block for Donor Site Pain in Stage I Microtia Reconstruction: A Pilot Study. Otolaryngol Head Neck Surg. 2016 May;154(5):898-901. doi: 10.1177/0194599816629395. Epub 2016 Feb 23. PMID 26908556
- [Derived] Wei S, Ye J, Lei C, Huang Q, Lin B, Su X, Zheng H, Shan X, Wang B, Wang M. Abdominal muscles infiltration analgesia for donor-site pain in autologous ear reconstruction: A randomized controlled clinical trial. J Plast Reconstr Aesthet Surg. 2024 Dec;99:38-46. doi: 10.1016/j.bjps.2024.09.019. Epub 2024 Sep 20. PMID 39342766